CLINICAL TRIAL: NCT02677246
Title: Phase 1 Trial of Denosumab for Prevention of Bone Complications After Allogenic Hematopoietic Stem Cell Transplantation in Children
Brief Title: Denosumab for Prevention of Bone Complications After Bone Marrow Transplantation in Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Pierre Teira, MD, MD, MSc, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSJ001
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Disorder Related to Bone Marrow Transplantation
Keywords: Bone marrow transplantation; Children; Bone complications; Denosumab.
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Denosumab (Experimental): Phase 1, 3+3 design with inter-patient dose escalation from 1mg/kg/dose to 2mg/kg/dose, and possibility of a dose de-escalation of 0.5mg/kg/dose, A modification of 3+3 design is implemented to take into account the achievement of bone resorption blockade by Denosumab. CTX is a biologic marker of bone resorption. Provided a decrease of CTX blood level will be observed under the lower limit (2,5th percentile) for age and sex, or under 20% of the pre-treatment level, there will be no reason to continue escalating the dose. This modified 3+3 design prevents exposure of children to dose escalations that would not be needed regarding the medical and biological aims of this trial.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Denosumab, one sub-cutaneous infusion, given within 2 weeks after engraftment defined as neutrophils > 0,5x10(9)/L and chimerism ≥ 10% of donor origin.
  Before starting Denosumab several requirements have to be met: 1) Calcemia and Phosphatemia in the normal ranges, 2) adequate Calcium and Vitamin D intakes according to age.
  Biological activity of Denosumab measured by CTX blood level, expected to last for 4 to 6 months after one infusion.
  Possibility of subsequent infusions at the same dose level, every 5 to 6 months, for patient remaining on corticotherapy, provided no DLT occurred and provided CTX blood level decreased under the required threshold, after the previous infusions of Denosumab

SUMMARY:
Children treated by bone marrow transplantation (BMT) experience bone toxicity. Those bone damages are caused by both a decrease of bone formation and an increase of bone destruction after BMT.For long term survivors, bone complications are major determinants of impaired quality of life. No standard treatment currently exists to prevent those bone injuries. Denosumab is a treatment which specifically blocks bone destruction for 4 to 6 months in adults. This trial will study whether it is safe to prescribe Denosumab to children after BMT in the aim of preventing bone complications.

DETAILED DESCRIPTION:
Participant will receive one subcutaneous dose of Denosumab within 2 weeks after confirmation of bone marrow engraftment. The dose of treatment will be escalated between participants. Denosumab is supposed to be effective for several months (4 to 6 months). The biologic activity of Denosumab will be followed by the measure in the blood of a biomarker of bone destruction called CTX. This biomarker is supposed to decrease after Denosumab infusion, reflecting the blockade of bone destruction by the treatment. Bone density will be assessed by a radiologic test named DXA which a standard test. All blood and radiologic tests mandated by the study will be done at the same time as standard follow-up after bone marrow transplant. Thus, participants will not have extra visits at the outpatient clinic, or extra blood punctures, for the specific purpose of the study. Participants will be followed for 36 months after bone marrow transplantation.For experiencing graft versus host disease, a second dose of Denosumab will be allowed, followed by subsequent doses evry 4 to 6 months till a maximum of 4 doses within 24months after bone marrow transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 2 year to 21 years
* Allogenic hematopoietic stem cell transplantation (allo-HSCT) planned within 1 month.
* Informed consent signed by participant more than 18 year old, or parents or his/her legal guardian
* Teeth examination by a dentist in order to rule out or to treat latent teeth infections before allo-HSCT

Exclusion Criteria:

* Refusal of signing informed consent
* Prior inclusion in another therapeutic trial with a time elapsed from the last research drug dose to Denosumab, shorter than 7 half-lifes of the research drug
* Osteopetrosis
* Bisphosphonates treatment within 12 months before entering the trial
* Tooth infection not treated before allo-HSCT
* Child-bearing and breastfeeding women

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerable Dose (MTD) | MTD will be definitively established at 6 months after the last patient has been entered into the study. Given the anticipated rate of accrual, the primary outcome measure should be determined within 2 years after opening the study.
  The MTD is defined as:
  * the maximum dose level at which 0 to 1 out of 6 patients experience dose-limiting toxicity (DLT) and above which 2 or more patients encounter DLT.
  * or the dose of Denosumab necessary for blocking bone resorption for at least 4 months in 6 consecutive patients, if dose limiting toxicities are not observed

SECONDARY OUTCOMES:
Evolution of CTX (a biological marker of bone resorption) level in blood | Dosage before transplantation, before beginning Denosumab, then monthly till 6 months, then at 12 months, 18 months, 24 and 36 months after starting Denosumab
  Duration of CTX level in blood on Denosumab treatment under the lower limit for age and sex, or less than 20% of the value before starting the conditioning regimen
Evolution of P1NP (a biological marker of bone synthesis) level in blood | Dosage before transplantation and before beginning Denosumab, then monthly till 6 months, then at 9 months, 12 months, 18 months, 24 months and 36 months after starting Denosumab
  Level of P1NP in blood at each time point of follow-up
Osteonecrosis (apart from jaw osteonecrosis) | At 1 year, 2 years and 3 years after bone marrow transplantation
  Cumulative Incidence of osteonecrosis based on clinical diagnosis at each time point of follow-up
Fracture | At 1 year, 2 years and 3 years after bone marrow transplantation
  Cumulative Incidence of fracture based on clinical diagnosis at each time point of follow-up
Bone Mineral Density (BMD) | Before bone marrow transplantation, then 6 months, 12 months, 24 months and 36 months after starting Denosumab
  BMD is measured by a routine radiologic test named dual energy X-ray (DXA) allowing to establish the Z score of BMD
Growth height evolution according to standardized World Health Organization growth charts for Canada | Measurement every 6 months till 24 months after entering the study, then yearly till 21 years of age.
  Evolution of growth height will be described as :
  * change in percentile between percentile of height before transplantation and percentile of height along time at each time point of follow-up
  * final height at the end of growth or at last follow-up
Dose Limiting toxicity (DLT) | Assessment every month till 6 months after bone marrow transplantation. For each dose level ,DLT will be established at 6 months after bone marrow transplantation of the 3rd participant entered into the cohort.
  Grade 3 to 5 toxicities probably or definitively related to Denosumab, if MTD is reach before a blockade of bone resorption is observed.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Teira, MD, Principal Investigator — St. Justine's Hospital
Locations (1):
- St. Justine 's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No